CLINICAL TRIAL: NCT05575011
Title: A Randomized, Blinded, Placebo-Controlled, Phase 1 Single Ascending Dose Study in Healthy Adult Male Volunteers and an Open-Label Multiple Ascending Dose Study With Long-Term Extension in Pediatric SMA Participants Previously Treated With Onasemnogene Abeparvovec (Zolgensma™) to Evaluate the Safety, Tolerability, and Pharmacokinetics of BIIB115
Brief Title: A Study to Learn About the Safety of BIIB115 Injections and How BIIB115 is Processed in the Bodies of Healthy Adult Male Volunteers and of Pediatric Participants With Spinal Muscular Atrophy Who Previously Took Onasemnogene Abeparvovec
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 277HV101; 2022-000956-12 (EudraCT Number); 2023-505643-39 (Other: EU CTIS Number)
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteer; Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: Sequential for Parts A, B, and B LTE parallel for Cohorts 1-4 within Part A, parallel for Cohorts 5-6 within Part B
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded for Part A and open-label for Part B of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A: Cohort 1: BIIB115 Dose 1 (Experimental): Participants will receive a single dose of BIIB115, Dose 1, via IT bolus injection, on Day 1.
  Interventions: Drug: BIIB115
- Part A: Cohort 2: BIIB115 Dose 2 (Experimental): Participants will receive a single dose of BIIB115, Dose 2, via IT bolus injection, on Day 1.
  Interventions: Drug: BIIB115
- Part A: Cohort 3:BIIB115 Dose 3 (Experimental): Participants will receive a single dose of BIIB115, Dose 3, via IT bolus injection, on Day 1.
  Interventions: Drug: BIIB115
- Part A: Cohort 4: BIIB115 Dose 4 (Experimental): Participants will receive a single dose of BIIB115, Dose 4, via IT bolus injection, on Day 1.
  Interventions: Drug: BIIB115
- Part A: Cohorts 1-4: BIIB115-Matching Placebo (Placebo Comparator): Participants will receive a single dose of BIIB115-matching placebo, via IT bolus injection, on Day 1.
  Interventions: Drug: BIIB115-Matching Placebo
- Part B: Cohort 5: BIIB115 Dose 3 (Experimental): Pediatric SMA participants previously treated with onasemnogene abeparvovec will receive two doses of BIIB115, Dose 3, via IT bolus injection at two separate time points.
  Interventions: Drug: BIIB115
- Part B: Cohort 6: BIIB115 Dose 4 (Experimental): Pediatric SMA participants previously treated with onasemnogene abeparvovec will receive two doses of BIIB115, Dose 4, via IT bolus injectionat two separate time points.
  Interventions: Drug: BIIB115
- Part B: Long Term Extension (LTE): BIIB115 Dose 4 (Experimental): Pediatric SMA participants previously treated with onasemnogene abeparvovec who have completed Part B and are eligible will receive five doses of BIIB115, Dose 4, via IT bolus injection at separate time points for up to 60-month duration.
  Interventions: Drug: BIIB115

INTERVENTIONS:
Drug: BIIB115 — Administered as specified in the treatment arm
  Arms: Part A: Cohort 1: BIIB115 Dose 1; Part A: Cohort 2: BIIB115 Dose 2; Part A: Cohort 3:BIIB115 Dose 3; Part A: Cohort 4: BIIB115 Dose 4; Part B: Cohort 5: BIIB115 Dose 3; Part B: Cohort 6: BIIB115 Dose 4; Part B: Long Term Extension (LTE): BIIB115 Dose 4
Drug: BIIB115-Matching Placebo — Administered as specified in the treatment arm
  Arms: Part A: Cohorts 1-4: BIIB115-Matching Placebo

SUMMARY:
In this study, researchers will learn about a study drug called BIIB115 in healthy adult male volunteers and in participants with spinal muscular atrophy (SMA). This study will focus on children with SMA.

The main objective of the study is to learn about the safety of BIIB115 and how participants respond to different doses of BIIB115. The main question researchers want to answer is:

• How many participants have adverse events and serious adverse events during the study?

Adverse events are unwanted health problems that may or may not be caused by the study drug.

Researchers will also learn about how the body processes BIIB115. They will do this by measuring the levels of BIIB115 in both the blood and the cerebrospinal fluid, also known as the CSF. This is the fluid around the brain and spinal cord.

The study will be split into 2 parts - Part A and Part B.

During Part A:

* After screening, healthy volunteers will be randomly placed into 1 of 4 groups to receive either BIIB115 or a placebo. A placebo looks like the study drug but contains no real medicine.
* Participants will receive a single dose of either BIIB115 or the placebo as an injection directly into the spinal canal on Day 1.
* Neither the researchers nor the participants will know if the participants will receive BIIB115 or the placebo.
* The Part A treatment and follow-up period will last for 13 months.
* Participants will have up to 6 clinic visits and 4 phone calls.

During Part B:

* After screening, children with SMA will be placed into 1 of 2 groups to receive BIIB115.
* The doses of each group will be decided based on the results of Part A.
* Both researchers and participants will know they are receiving BIIB115.
* Participants will first receive 2 total doses of BIIB115 given at 2 different times.
* The Part B treatment and follow-up period will last for 24 months.
* Participants will have up to 14 clinic visits and 6 phone calls.

Part B Long-Term Extension:

* After completing the 25 months in Part B, participants may move onto the long-term extension (LTE).
* They will receive 5 more doses of BIIB115 at different times.
* The Part B LTE treatment and follow-up will last for 60 months.
* Participants will have up to 12 more clinic visits and 19 phone calls. In both Part A and Part B, participants will stay in the clinic for 24 hours after each dose so that researchers can check on their health. This 24-hour stay will not be required for the Part B LTE period.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the safety and tolerability of BIIB115 administered via intrathecal (IT) bolus injection to healthy participants in Part A, pediatric participants with spinal muscular atrophy who have previously received onasemnogene abeparvovec in Part B, and to participants who complete Part B in Part B LTE. The secondary objectives of the study is to evaluate the pharmacokinetics (PK) of BIIB115 in Parts A, B, and B LTE.

ELIGIBILITY:
Key Inclusion Criteria:

Part A:

* Male healthy participants aged 18 to 55 years, inclusive
* Have a body mass index of 18 to 30 kilograms per meter square (kg/m^2), inclusive
* Must be in good health as determined by the investigator, based on medical history and screening evaluations

Part B:

* Age 0.5 to 12 years old, inclusive, at the time of informed consent
* Weight ≥7 kg at the time of informed consent
* Genetic diagnosis of SMA (5q SMA homozygous survival motor neuron 1 (SMN1) gene deletion or mutation or compound heterozygous mutation)
* Survival motor neuron 2 (SMN2) copy number ≥1
* Must have received intravenous (IV) onasemnogene abeparvovec per the approved label or per guidelines including the steroid regimen and monitoring specified therein
* Treatment with onasemnogene abeparvovec ≥180 days prior to first BIIB115 dose
* Potential for improvement due to suboptimal clinical status secondary to SMA, as determined by the Investigator

Part B LTE

* Completion of the assessments in Part B
* Meets age-appropriate institutional criteria for use of anesthesia/sedation, if use is planned for study procedures (as assessed by the Investigator and either anesthesiologist or pulmonologist).

Key Exclusion Criteria:

Part A:

* Any reason, anatomical or otherwise (including abnormal hematology/coagulation), that presents increase of risk of complication from multiple lumbar puncture (LP) procedures required for dosing and CSF collection, per the investigator discretion
* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator
* Chronic, recurrent, or serious infection, as determined by the investigator, within 90 days prior to screening or between screening and Day -1
* Current enrollment or a plan to enroll in any interventional clinical study of a drug, biologic, or device, in which an investigational treatment or approved therapy for investigational use is administered within 3 months (or 5 half-lives of the agent, whichever is longer) prior to randomization

Part B:

* Severe or serious AEs related to onasemnogene abeparvovec therapy that are ongoing during Screening
* Interval of <180 days between onasemnogene abeparvovec therapy and first BIIB115 dose
* Ongoing steroid treatment following onasemnogene abeparvovec at time of screening
* History of drug induced liver injury or liver failure per Hy's law definition
* History of thrombotic micrangiopathy
* Treatment with any SMN2-splicing modifier (nusinersen or risdiplam) after receiving onasemnogene abeparvovec. Treatment with nusinersen <12 months from the first dose of BIIB115.
* Any reason, anatomical or otherwise (including abnormal hematology/coagulation), that presents increase of risk of complication from the LP procedures, CSF circulation, or safety assessments, including a history of hydrocephalus or implanted shunt for CSF drainage.
* Permanent ventilation, defined as tracheostomy or ≥16 hours ventilation /day continuously for >21 days in the absence of an acute reversible event

Part B LTE:

* Any new condition or worsening of an existing condition that, according to the Investigator, would make the participant unsuitable for inclusion, could interfere with the assessment of safety, or would compromise the ability of the participant to undergo study procedures.
* Clinically significant abnormalities in hematology, blood chemistry parameters, or electrocardiograms (ECGs) prior to first LTE visit that would make the participant unsuitable for inclusion as assessed by the Investigator.
* Treatment with an approved SMN2-splicing modifier (nusinersen or risdiplam).

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 6 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2031-11-14 (Estimated); Study Completion 2031-11-14 (Estimated)

PRIMARY OUTCOMES:
Parts A, B, and B Long Term Extension (LTE): Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Part A: Up to Day 393, Part B: Up to Day 720; Part B LTE: Up to Day 2520
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.

SECONDARY OUTCOMES:
Parts A, B, and B LTE: Concentration of BIIB115 in Cerebral Spinal Fluid (CSF) | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720; Part B LTE: Day 720 to Day 2520
Part A: Terminal Elimination Half-Life (t½) of BIIB115 in CSF | Day 1 to Day 180
Parts A, B, and B LTE: Concentration of BIIB115 in Serum | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720; Part B LTE: Day 720 to Day 2520
Parts A and B: Terminal Elimination Half-Life (t½) of BIIB115 in Serum | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720
Parts A and B: Area Under the Concentration-Time Curve from Time 0 to Last Measurable Concentration (AUC0-last) of BIIB115 in Serum | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720
Parts A and B: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUCinf) of BIIB115 in Serum | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720
Parts A and B: Maximum Observed Concentration (Cmax) of BIIB115 in Serum | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720
Parts A and B: Time to Reach Maximum Observed Concentration (Tmax) of BIIB115 in Serum | Part A: Day 1 to Day 180, Part B: Day 1 to Day 720

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (17):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Children's Hospital of Eastern Ontario, Ontario, Canada
- Hôpital Armand Trousseau, Paris, France
- Germany (3):
  - Universitatsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Heidelberg, Heidelberg
- Italy (2):
  - Fondazione Serena Onlus - Centro Clinico Nemo, Milan
  - Pediatric Neurology Unit, Catholic University, Rome
- Netherlands (2):
  - Centre For Human Drug Research, Leiden
  - UMC Utrecht, Utrecht
- Poland (3):
  - Instytut Centrum Zdrowia Matki Polki Dept of Neurology, Lodz
  - PRATIA S.A. MTZ Clinical Research Powered by Pratia, Warsaw
  - Instytut "Pomnik - Centrum Zdrowia Dziecka, Warsaw
- South Korea (2):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, Bloomsbury
  - Sheffield Childrens Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/